CLINICAL TRIAL: NCT00725101
Title: Real World Examination of Fibromyalgia: Longitudinal Evaluation of Costs and Treatments (The REFLECTIONS Study)
Brief Title: Fibromyalgia Health Outcome Study on Cost of Treatments
Acronym: REFLECTIONS
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 11540; F1J-MC-B020 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fibromyalgia (FM) Participants: FM participants starting any new pharmacologic FM agent.
  Interventions: Drug: Treatment for Fibromyalgia

INTERVENTIONS:
Drug: Treatment for Fibromyalgia — FM participants starting any new pharmacologic FM agent.

SUMMARY:
The Real World Examination of Fibromyalgia: Longitudinal Evaluation of Costs and Treatments (REFLECTIONS) Study is a 12-month, prospective observational study that will be utilized in approximately 58 care settings in the United States (US) and Puerto Rico. It is designed to examine treatment patterns and health outcomes of adult participants diagnosed by their physician with fibromyalgia (FM) and who are starting any "new pharmacologic agent" for FM.

The primary benefit of this study is enhanced understanding of the disease state of FM and the role that pharmacologic treatment plays, which may help to optimize management of FM. This study will address current gaps in a rapidly growing body of literature on FM.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for fibromyalgia (FM) in the opinion of the investigator
* Must be prescribed a 'new' treatment for FM
* Male and female participants at least 18 years of age
* Willing to complete the Informed Consent Document (ICD) and any other required forms to be eligible for study participation
* Currently under the care of the participating physician
* Cognitively able to understand and complete participant self-rated scales in English or Spanish via computer-assisted telephone interview (CATI)
* Available for 12 months to participate in the study

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Are Lilly employees
* Are Terminally ill
* Currently participating in other research studies or if beginning a research study while participating in this study
* Unable to respond via telephone for CATI
* Incompetent for interview as deemed by the participating physician
* Unwilling to provide written ICD or other required forms to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple care centers
Sampling Method: Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (58):
- United States (49):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Blue Ridge, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Snellville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nampa, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fishers, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Towson, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Plains, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dover, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Brunswick, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medford, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schenectady, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boone, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minot, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Findlay, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Reading, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flower Mound, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garland, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Prairie, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirkland, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beckley, West Virginia
- Puerto Rico (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cidra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Humacao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayagüez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Isabel

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fibromyalgia (FM) Participants
Started | 1700
Completed | 1205
Not Completed | 495
Not completed — Death | 3
Not completed — Lost to Follow-up | 353
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 127
Not completed — not specified/no reason given | 11

BASELINE CHARACTERISTICS:
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1700
Age Continuous [Mean (Standard Deviation); unit: years] | 50.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1601
  Male | 99
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1391
  Hispanic | 209
  Other | 100
Region of Enrollment [Number; unit: participants]
  United States | 1539
  Puerto Rico | 161
Number of Unique Baseline Medications Taken for Fibromyalgia (FM; Newly-Initiated and Continuing) [Number; unit: unique baseline medications] | 181
Mean Number of Concurrent Baseline Medications Taken for Fibromyalgia (FM) [Mean (Standard Deviation); unit: concurrent baseline medications] | 2.6 (1.2)
Brief Pain Inventory-Severity (BPI-S) Average Subscale Score [Mean (Standard Deviation); unit: units on a scale] — BPI-S measures self-reported severity of pain. Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine) for each question assessing worst pain, least pain, and average pain in the past 24 hours, and current pain.
  units on a scale | 5.5 (1.8)
Brief Pain Inventory-Interference (BPI-I) Average Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Average BPI-I measures self-reported degree of pain interference on function. Interference scores range from 0 (does not interfere) to 10 (completely interferes) for each question assessing interference of pain within the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
  units on a scale | 6.1 (2.2)
Fibromyalgia Impact Questionnaire (FIQ) [Mean (Standard Deviation); unit: units on a scale] — FIQ measures self-reported fibromyalgia (FM) status, progress, and outcomes over past week. FIQ has 20 items: Items 1-11 measure physical functioning (each rated on 4-point Likert-type scale); Items 12 + 13 measure number (no.) of days participant felt well and no. of days participant felt unable to work due to FM symptoms. Items 14-20 are numerical, 11-point Likert-type scales (marked in 10-millimeter [mm] increments) rating work difficulty, pain intensity, fatigue, morning tiredness, stiffness, anxiety, and depression. Total scores range from 0 to 80; Higher score=greater negative impact.
  units on a scale | 54.4 (13.7)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: units on a scale] — SDS is a self-rated measurement of disability across 3 domains: work/school, social life, and family life/home responsibilities. Participant marks along the line from 0 (not at all) to 10 (extremely disrupted), the number that best represents how much each area is disrupted by fibromyalgia symptoms.
  units on a scale | 18.3 (7.6)
Opioid Use [Number; unit: participants]
  No | 1288
  Yes | 412
Nonsteroidal Anti-Inflammatory Drug (NSAID) Use [Number; unit: participants]
  No | 1245
  Yes | 455
Main Reasons for Discontinuing Medications Before Starting Fibromyalgia (FM) Treatment at Baseline [Number; unit: participants] — Physicians reported the single, main reason for a participant to discontinue a medication during the Baseline visit. The number of participants included those who discontinued medication before starting fibromyalgia treatment at Baseline.
  participants
    Felt better | 6
    Did not help | 332
    Adverse events | 81
    Too costly | 14
    Other | 59

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Medications Taken for Fibromyalgia (FM) Over 12 Months
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who took part in all follow-up interviews.
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1073
medications | 5.2 (2.1)

2. Primary Outcome: Odds Ratio From Stepwise Logistic Regression Model of Baseline Medication Use for Fibromyalgia (FM): Duloxetine, Pregabalin, or Milnacipran Versus Any Other Medication
Description: Significant variables included in the final model were age over 65, physician gender and specialty, use of opioids (excluding tramadol), use of non-steroidal anti-inflammatory drugs (NSAIDs), and number of medications.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had non-missing covariates used in logistic regression.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1275
odds ratio
  Age over 65 | 0.535 [0.338 to 0.845]
  Female physician | 1.665 [1.192 to 2.325]
  Rheumatology versus Primary Care Physician (PCP) | 2.662 [1.864 to 3.802]
  Other specialty versus PCP | 2.671 [1.758 to 4.060]
  Use of opioids | 0.667 [0.498 to 0.893]
  Use of NSAIDs | 0.447 [0.337 to 0.594]
  Number of baseline medications taken | 1.394 [1.247 to 1.558]
Statistical Analysis 1: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.0074, Regression, Logistic — P-value for age over 65
Statistical Analysis 2: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.0028, Regression, Logistic — P-value for female physicians
Statistical Analysis 3: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — P-value for Rheumatology versus PCP
Statistical Analysis 4: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — P-value for other specialty versus PCP
Statistical Analysis 5: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.0064, Regression, Logistic — P-value for use of opioids
Statistical Analysis 6: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — P-value for use of NSAIDs
Statistical Analysis 7: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — P-value for number of medications participants were taking

3. Primary Outcome: Odds Ratios From Stepwise Logistic Regression Model of Longitudinal Adherence to Duloxetine Treatment for Fibromyalgia (FM) Over 12 Months: Generalized Anxiety Disorder-7 (GAD-7) Score, Pregabalin Use, and Non-Steroidal Anti-Inflammatory Drug (NSAID) Use
Description: Significant variables included in the final model were pregabalin use, NSAID use, and GAD-7 (7-item, self-reported measurement of GAD severity [not at all severe, severe for several days, severe for more than half the days, severe nearly every day]; Total score=sum of all 7 items; ranges from 0 to 21; Higher score=greater level of anxiety). Odds ratios were based on medication possession ratio (MPR) ≥0.8 for pregabalin and NSAID use among duloxetine initiators at Baseline; MPR=total supply days/total number of days in 12-month study period.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had non-missing covariates used in logistic regression.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 212
odds ratio
  GAD-7 | 1.06 [1.01 to 1.12]
  Pregabalin use | 2.69 [1.16 to 6.22]
  NSAID use | 2.25 [1.00 to 5.08]
Statistical Analysis 1: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.026, Regression, Logistic — P-value for GAD-7 score
Statistical Analysis 2: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.021, Regression, Logistic — P-value for pregabalin use
Statistical Analysis 3: Comparison: Fibromyalgia (FM) Participants; Test type: Superiority or Other; p = 0.050, Regression, Logistic — P-value for NSAID use

4. Secondary Outcome: Reasons for Discontinuing Medications for Fibromyalgia (FM) During the Study
Description: Participants were allowed to select multiple reasons for discontinuing treatment. During the 12-month period post-baseline, a participant could possibly discontinue more than 1 medication, or discontinue the same medication more than once. A reason for discontinuation was given each time a participant stopped taking a medication.
Time Frame: Baseline through 12 months
Population: The analysis population included participants who reported discontinuing medication at least once during the 12-month period post-baseline.
Measure: Number; unit: participants
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 978
participants
  Felt better | 49
  Did not help | 637
  Adverse events | 731
  Too costly | 121
  Other | 458
  No reason provided | 116

5. Secondary Outcome: Percentage of Participants Who Discontinued Opioids
Time Frame: Baseline through 12 months
Population: The analysis population included participants who were using opioids at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 412
percentage of participants
  Discontinued opioid use by 3 months of treatment | 11.9
  Discontinued opioid use by 6 months of treatment | 15.3
  Discontinued opioid use by 12 months of treatment | 22.0

6. Secondary Outcome: Hazard Ratios for Factors Associated With Discontinued Opioid Use
Description: Factors significantly associated with discontinuation of opioid use were participant age, Brief Pain Inventory-Interference (BPI-I) score, and Patient Health Questionnaire for somatic symptoms (PHQ-15) score.
Time Frame: Baseline through 12 months
Population: The analysis population included participants who were using opioids at Baseline.
Measure: Number; unit: hazard ratio
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 325
hazard ratio
  Age: younger more likely to discontinue | 0.97
  BPI-I: higher baseline score=more likely | 1.57
  PHQ-15: lower baseline score=more likely | 0.93

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Interference (BPI-I) Average Subscale Score at 12 Months
Description: Average BPI-I measures self-reported degree of pain interference on function. Interference scores range from 0 (does not interfere) to 10 (completely interferes) for each question assessing interference of pain within past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: Baseline, 12 months
Population: The analysis population included participants who had non-missing BPI-I scores at Baseline and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1202
units on a scale | -0.66 (2.12)

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Severity (BPI-S) Average Subscale Score at 12 Months
Description: BPI-S measures self-reported severity of pain. Severity scores range from 0 (no pain) to 10 (severe pain) for each question assessing worst pain, least pain, and average pain in past 24 hours, and current pain.
Time Frame: Baseline, 12 months
Population: The analysis population included participants who had non-missing BPI-S scores at Baseline and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1172
units on a scale | -0.33 (1.72)

9. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Total Score at 12 Months
Description: FIQ measures self-reported fibromyalgia (FM) status, progress, and outcomes over past week. FIQ comprises 20 items: Items 1-11 measure physical functioning (each rated on 4-point Likert-type scale); Items 12 + 13 measure number (no.) of days participant felt well and no. of days participant felt unable to work due to FM symptoms. Items 14-20 are numerical, 11-point Likert-type scales (marked in 10-millimeter [mm] increments) rating work difficulty, pain intensity, fatigue, morning tiredness, stiffness, anxiety, and depression. Total scores range from 0-80; Higher score=greater negative impact.
Time Frame: Baseline, 12 months
Population: The analysis population included enrolled participants who had non-missing FIQ scores at Baseline and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1182
units on a scale | -3.81 (13.47)

10. Secondary Outcome: Change From Baseline in Sheehan Disability Score (SDS) Total Score at 12 Months
Description: The SDS is completed by the participant and assesses the effect of the participant's symptoms on work/social/family life. Total scores range from 0 to 30; Higher score=greater disruption in the participant's work/social/family life.
Time Frame: Baseline, 12 months
Population: The analysis population included enrolled participants who had non-missing SDS scores at Baseline and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1180
units on a scale | -2.28 (7.26)

11. Secondary Outcome: Number of Outpatient Visits Due to Fibromyalgia (FM)
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit. The number of participants actually used in analyses were less than 1700 because some had missing outpatient visit values.
Measure: Mean (Standard Deviation); unit: outpatient visits
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1600
outpatient visits | 21.2 (28.6)

12. Secondary Outcome: Number of Emergency Room (ER) Visits Due to Fibromyalgia (FM)
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit. The number of participants actually used in analyses were less than 1700 because some had missing ER visit values.
Measure: Mean (Standard Deviation); unit: ER visits
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1598
ER visits | 0.9 (2.5)

13. Secondary Outcome: Number of Days of Partial Care for Fibromyalgia (FM) Participants
Description: Partial (day or night) care included day care, day nursing home, and partial hospitalization.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1600
days
  Partial day care | 1.2 (8.1)
  Partial night care | 0.6 (3.9)

14. Secondary Outcome: Number of Days of Caregiver Burden Due to Fibromyalgia (FM; Family Missed Paid Work and Used a Paid Caregiver)
Description: Caregiver burden was described as the number of days family members missed paid work and used a paid caregiver (for example, home healthcare nurse) to care for the participant with FM.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1600
days
  Days family missed paid work | 2.7 (12.2)
  Days family used paid caregiver | 2.7 (17.6)

15. Secondary Outcome: Number of Days of Caregiver Burden Due to Fibromyalgia (FM; Family Used an Unpaid Caregiver)
Description: Caregiver burden was described as the number of days family members used an unpaid caregiver (family and friends) to care for the participant with FM.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1599
days | 36.4 (76.6)

16. Secondary Outcome: Number of Days Fibromyalgia (FM) Affected Participant Productivity (Stayed in Bed, Reduced Activity, and Received Disability Income)
Description: Participant productivity was described as the number of days the participant stayed in bed, had to reduce normal activity by half, and received disability income due to FM.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1600
days
  Days participant stayed in bed due to FM | 40.6 (58.2)
  Days participant reduced activity by at least half | 86.5 (76.3)
  Days participant received disability income | 98.2 (148.3)

17. Secondary Outcome: Number of Days Fibromyalgia (FM) Affected Participant Productivity (Missed Work)
Description: Participant productivity was described as the number of days a participant missed work due to FM.
Time Frame: Baseline through 12 months
Population: The analysis population included enrolled participants who had at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fibromyalgia (FM) Participants
Number analyzed (Participants) | 1590
days | 25.0 (56.1)

ADVERSE EVENTS:
Description: This observational study was not designed to collect or monitor safety data. To maintain non-interventional methods, per the protocol/study design, adverse events (AEs) were not collected, and physicians were instructed to handle AEs according to laws and regulations for US-marketed drugs.
Arm/Group | Fibromyalgia (FM) Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days